CLINICAL TRIAL: NCT06294249
Title: The Evaluation of Pain Severity in Flapless Dental Implant Placement Using Laser-induced Incisions: A Split Mouth Randomized Clinical Trial Study
Brief Title: Pain Severity in Flapless Dental Implant Placement Using Laser
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Tabrizi, DMD, Associate Professor of Oral and Maxillofacial Surgery, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20045125
Record Dates: First submitted 2024-01-22; First posted 2024-03-05 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Jaw, Edentulous, Partially
Keywords: Jaw, Edentulous, Partially; Pain Measurement; Laser Therapy; Dental Implants; Randomized Controlled Trial
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Laser-induced Incision (Experimental): The Biolase Epic 10 diode laser device (Biolase, USA) with 940 nm wavelength, 10 W of max output power, 20 KHz of pulse repetition rate, and continuous pulse mode was used.
  Interventions: Device: Laser-induced Incision; Procedure: Implant Placement
- Punch Incision (Active Comparator): The soft tissue Osstem punch (South Korea) was used.
  Interventions: Procedure: Punch Incision; Procedure: Implant Placement

INTERVENTIONS:
Device: Laser-induced Incision — On the treatment side, an incision was made on the crest of the alveolar soft tissue using the laser.
  Arms: Laser-induced Incision
Procedure: Punch Incision — On the control side, a punch incision was made on the crest of the alveolar soft tissue using using a punch.
  Arms: Punch Incision
Procedure: Implant Placement — Implant placement was done in both laser and punch arms. The drilling was performed based on the company (Straumman) protocol. On each side, a dental implant (Straumman SP, Basel, Switzerland) and healing abutment were placed. Patients were visited at 24, 48, 72 hours, and 7 days after insertion.

SUMMARY:
The goal of this split-mouth randomized clinical trial study was to investigate the effect of using a laser on pain and discomfort following flapless dental implant surgery. It was hypothesized that laser did not have any impact on post-op pain. Therefore, the study aimed to compare pain and discomfort following flapless dental implant surgeries with or without a laser.

ELIGIBILITY:
Inclusion Criteria:

1. Adult human subjects agreed to participate in the study and return on follow-up times
2. Subjects eligible for receiving dental implants
3. Subjects with an edentulous area in the posterior of the mandible bilaterally 3- Subjects with sufficient bone width and height (>5 mm width, and >10 mm height) at the implant sites
4. Subjects with sufficient keratinization tissue at the implant sites

Exclusion Criteria:

1. Subjects refused to return for follow-up or refused study enrollment.
2. Subjects with uncontrolled systemic diseases
3. Subjects younger than 18 years
4. Subjects receiving psychotropic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Patients were visited at 24, 48, 72 hours, and 7 days after insertion.
  Measured using the visual analogue scale (VAS): 0-3 mild pain, 4-6 moderate pain, and 7-10 sever pain.

CONTACTS AND LOCATIONS:
Overall Officials: +98-9125850829 Tabrizi, DMD, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- shiraz University of medical sciences, Shiraz, Fars, Iran